CLINICAL TRIAL: NCT02836197
Title: Communication About Uncertainty and Hope: A Randomized Controlled Trial Assessing the Efficacy of a Communication Skills Training Program for Physicians Caring for Cancer Patients
Brief Title: Randomized Controlled Trial Assessing the Efficacy of a Communication Skills Training Program
Acronym: CERTAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Collaborators: Université Libre de Bruxelles (Other); Université Catholique de Louvain (Other); Université de Liège (Other); Centre de Psycho-Oncologie (CPO) (Other)
Responsible Party: Principal Investigator, Yves Libert, Professor, Jules Bordet Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CERTAIN
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Physician Patient Relationship
Keywords: Uncertainty;hope;cancer;communication skills training;physicians

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group of 30 physicians will immediately attend the intervention communication skills training program (experimental group).For this experimental group, the first assessment will take place before the first training session and the second recording after the last session. This assessment involves the analyses of communicational, physiological and psychological variables recorded in the context of an encounter with a simulated advanced stage cancer patient.
  Interventions: Behavioral: Communication skills training
- Waiting-list group (No Intervention): This group of 30 physicians will attend the intervention communication skills training in a delayed manner (control group). For this control group, the first and the second recording will take place with a four-month interval. This assessment involves the analyses of communicational, physiological and psychological variables recorded in the context of an encounter with a simulated advanced stage cancer patient.

INTERVENTIONS:
Behavioral: Communication skills training — The general aim of the communication skills training program is to help physicians learn effective communication skills in contexts of high uncertainty. The training will last 30 hours, will be spread over 4 months. The training will be conducted by group of 3 subjects. The training will include mainly role-plays, theoretical information and modeling techniques. A training manual has been developed to increase content standardization and reduce potential group or trainee biases. The role-plays will be based on clinical cases brought up by the participants.
  Arms: Experimental group

SUMMARY:
Background: Although previous studies have reported the efficacy of communication skills training programs (CST), specific training addressing communication about uncertainty and hope in oncology has not yet been studied. This paper describes the study protocol of a randomized controlled trial assessing the efficacy of a CST program aimed at improving physician ability to communicate about uncertainty and hope in encounters with cancer patients.

Methods: Physician participants will be randomly assigned in groups (n = 3/group) to a 30-hour CST program (experimental group) or to a waiting list (control group). The training program will include learner-centered, skills-focused, practice-oriented techniques. Training efficacy is assessed in the context of an encounter with a simulated advanced stage cancer patient at baseline and after the CST for the experimental group, and after four months for the waiting-list group. Efficacy assessments will include communicational, psychological and physiological measures. Group-by-time effects will be analyzed using a generalized estimating equation (GEE). A power analysis indicated that a sample size of 60 (30 experimental and 30 control) participants will be sufficient to detect effects.

Discussion: The current study will aid in the development of effective CST programs to improve physician ability to communicate about uncertainty and hope in encounters with cancer patients.

DETAILED DESCRIPTION:
1. Aim of the trial A randomized longitudinal study assessing the efficacy of a CST program aimed at improving physician communication about uncertainty and hope with cancer patients will be conducted. Efficacy of the program will be assessed by the analysis of changes over time in physician communication skills and physician psychological and physiological health. These assessments will be performed in the context of an encounter with a simulated advanced-stage cancer patient.
2. Subjects Participants will be physicians that are specialists or residents, have a practice including cancer patients and speak French. The study was approved by a central ethics committee (Jules Bordet Institute, Cancer Center of the Université Libre de Bruxelles) and all participants will provide written informed consent.
3. Study Design Participating physicians will be randomly assigned to either the experimental group or the control group (Figure 1). After baseline assessment, participants in the experimental group will attend a 4-month training program followed by a post assessment. Participants in the control group will be placed on a training program waitlist after baseline assessment and will be reassessed four to five months later. The process of randomization after baseline will allow for a double-blind assessment at baseline.
4. CST Program 4.1. CST aims The aim of the CST is to improve the ability of physicians to communicate about uncertainty and hope with cancer patients.

   4.2. CST logistics The CST is a manualized program comprised of ten 3-hour sessions (30 hours) spread over four to five months. Each training group will include three physicians. The training will be conducted at locations and times choosen by the physicians within each group. The trainer of the experimental group will be an experienced facilitator who will conduct all training sessions (Y.L.). The training timetable will not include more than two 3-hours sessions in one day. Physicians will have the opportunity to register in groups of three or individually. In the latter case, physicians will be assigned to groups according to geographical proximity.

   4.3. CST Sessions The first session of the training program will include a general introduction to training and a modeling session. Sessions two to four will focus on appropriate communication skills for addressing uncertainty and hope according to a model detailed in a training manual. During sessions five to seven, participants will learn to transfer their newly-learned skills to clinical practice. Finally, during sessions eight to ten, skills learned during the training program will be consolidated.

   4.4. CST Program The CST program will include theoretical information giving about uncertainty and hope in cancer care (based on psychodynamics, cognitive-behavioral and systemic theories), modeling and role-playing.
   * Theoretical information giving The CST trainer will provide theoretical information on communication skills needed to address uncertainty and hope in encounters with cancer patients. These skills will focus on assessing patient expectations about the future and restructuring patient understandings with appropriate information when needed; and assessing patient hopes about the future and supporting those which are realistic [47]. All skills will be based on a collaborative and bidirectional communication process between physicians and patients on topics such as disease prognosis or expected and unexpected medical, psychological and social effects of cancer treatments. A specific algorithmic theoretical model has been designed to aid physicians in the implementation of these communication skills.
   * Modeling During the first CST session, physicians will observe a 16-minute video of a simulated interview in which the trainer acts as a physician communicating with a patient suffering from advanced cervical cancer. In the scenario, the patient has come for chemotherapy treatment and is requesting reassurance about treatment efficacy.

   The modeling session will empahsize three factors: 1) physician attitudes necessary to address uncertainty and hope, 2) patient's reactions to the discussion of uncertainty and hope and 3) the need to set up a safe and comfortable setting in which to model communication skills needed to address uncertainty and hope. After the video, physicians will be given one hour to debrief and react to the simulated interview.

   • Role-playing Throughout training, participants will be invited to participate in interactive role-playing with immediate and circular feed-backs [48]. Physicians will be asked to identify a clinical situation for the focus of the role-play situation. In session two to four, physicians will be asked to define a situation that would be highly uncomfortable in terms of uncertainty and hope management. In training sessions five to seven, physicians will be asked to identify clinical situations in which the transfer of learned communication skills would be difficult. Finally, in training sessions eight to ten, physicians will be asked to identify clinical situations during which the transfer of acquired skills would be uncomfortable.

   During role-play, the physician who reports the clinical situation will take on the role of the patient. This will allow role-play to be as realistic as possible. The small group context will promote an interactive session. During role-play, the "patient" will be exposed to the ways that he and his two colleagues are communicating in repeated rotations. During each rotation, the facilitator will suggest alternative strategies that were taught in the theoritical model and shown in the modeling video.

   • Transfering to clinical practice Each training session will start with a 15-minute summary of material learned since the beginning of the training program along with a debriefing from participants of attempts to transfer the learned skills to their clinical practice. Each training session will end with a 10-minute summary of the skills learned during the session, the difficulties that may have been encountered, and a proposal for the transfer of newly learned skills to future encounters with patients.
5. Assessment Procedure The performance status, disease status and communication skills among cancer patients vary widely and as such, the use of standardized encounters with simulated patients has been recommended to assess the efficacy of CST programs designed for healthcare professionals [49]. The assessment procedure for the current study will involve the video recording of an encounter between the participating physician and a simulated advanced stage cancer patient. Participating physicians will be assessed individually. An investigator, not involved in the training program, will present each subject with questionnaires. The assessment procedure (Figure 2) will include 7 steps: (1) continuous monitoring of heart rate, (2) relaxation exercise, (3) administration of questionnaires, (4) review of the simulated cancer patient medical chart, (5) administration of the second set of questionnaires, (6) encounter with the simulated cancer patient and (7) final set of questionnaires. Perceived stress will be measured seven times throughout the assessment procedure.

5.1. Simulated Patient Encounter The simulated patient case was written by an oncologist and a psycho-oncologist at the medical oncology unit and the psycho-oncology clinic at the Jules Bordet Institute, Cancer Center of the Université Libre de Bruxelles. The simulated patient case was developed to increase physician uncertainty about predefined medico-psycho-social components and available evidence-based treatments. The simulated patient is a 36-year-old woman with advanced cancer. She is facing a third recurrence (hepatic metastasis) of a breast cancer that had previously been treated with surgery, hormone therapy, radiation therapy and chemotherapy. She has agreed to start a new chemotherapy treatment. The scenario specifies that the patient has requested a meeting with a physician to help her cope with her treatment decision. Participants will be instructed to address and respond to the concerns of the simulated patient and to take the time they need for doing that. The simulated patient will be played by an actress experienced in simulated patient encounters and will be trained to maintain a standardized script and behavior. Regular feedback sessions will be held to help the actress maintain reproducibility [50]. The simulated patient encounters will take place at the Communication Laboratory (LabComm) of the Centre de Psycho-Oncologie (Brussels, Belgium).

5.2. Psychological Assessments Participating physicians will be asked to complete a set of psychological questionnaires prior to reading the patient medical file. Data on socioprofessional characteristics, practices in oncology and sense of mastery of the communication skills needed to address uncertainty and hope with cancer patients will be collected. A second set of psychological questionnaires administered immediately prior to the encounter with the simulated patient will gather information on the perceived realism of the medical chart of the simulated patient, agreement with the treatment decision, outcome expectancies on the medical, psychological and social status of the simulated patient, perceived uncertainty and hope regarding the medical, psychological and social outcomes of the simulated patient, and psychological reactions to uncertainty regarding the medical, psychological and social outcomes of the simulated patient. Finally, a third set of psychological questionnaires will be administered immediately after meeting with the simulated patient. These questions will pertain to agreement with the treatment decision, satisfaction regarding the encounter with the simulated patient, and the sense of mastery regarding the communication skills used to address uncertainty and hope with the simulated patient. These psychological questionnaires will allow the assessment of predictors and correlates of communication skill learning used to address uncertainty and hope with the simulated patient.

5.3. Communication Assessments The encounter with the simulated patient will be video recorded and transcribed. Physician communication skills will be analyzed using three tools. The French communication content analysis software, LaComm (Centre de Psycho-Oncologie, Brussels, Belgium; http://www.lacomm.be/) analyzes verbal communication (in medicine in general and in oncology in particular) and identifies turns of speech and the type and content of speech. The explanation of how this software works has been detailed in previous publications [42, 51]. The Multidimensional analysis of Patient Outcome Predictions (MD.POP) is a reliable tool used to measure verbal expressions that address the clinical future of a patient during medical encounters. This coding system allows one to manually identify, code, and score detailed verbal content from a medical encounter transcript that addresses a patient's clinical future. The detailed MD.POP codebook is available upon request. Finally, a specific interaction-process analysis system assessing communication skills addressing hope and uncertainty will be developed for the study [52].

5.4. Physiological Assessments Throughout all assessment procedures, physician heart rate will be monitored to assess the impact of the training program on the physiological arousal associated with communication about uncertainty and hope with the simulated patient. This assessment procedure has previously been used to measure the effect of CST on the physiological arousal of residents breaking bad news in a simulated task [53].

5.5. Statistical Analyses The primary outcome of the current study is the physicians' increased communication performance after training during this encounter. A power analysis has been performed, based on a previous longitudinal study assessing physicians' communication performance composite score in an encounter with a simulated advanced-stage cancer patient (Mean = 26; SD = 8) [54]. This power analysis was conducted considering 4 independent conditions according to the time (time 1 versus time 2) and the group (experimental versus control group). As there is no previous study assessing the efficacy of an intensive communication skills training program on physicians' communication about uncertainty and hope, it was hypothesized that physicians in the control group will maintain a stable performance score from time 1 to time 2. It was also hypothesized that physicians in the experimental group will improve their performance score by 20% from time 1 to time 2. Sample size calculation has been based on an 80% power, a one-sided α = 0.05 t-test and an effect size of 0.65. Considering this power analysis, 60 evaluable physicians are therefore needed for the efficacy assessment. Considering a drop-out rate of 20%, 12 physicians should be moreover recruited (72 physicians in total). It should be recalled at this level that one trainer only will conduct the training of the experimental group. Secondary, to assess also the CST program efficacy, group-by-time effects will be performed using generalized estimating equation (GEE) on psychological, physiological and communicational assessments performed during the encounter with the simulated patient.

BIBLIOGRAPHY

1. Snyder, C.R., et al., The Will and the Ways: Development and Validation of an Individual-Differences Measure of Hope. Journal of Personality and Social Psychology, 1991. 60(4): p. 570-585.
2. de Figueiredo, M.N., et al., ComOn Coaching: Study protocol of a randomized controlled trial to assess the effect of a varied number of coaching sessions on transfer into clinical practice following communication skills training. BMC cancer, 2015. 15(1): p. 503.
3. Razavi, D., et al., Testing health care professionals' communication skills: The usefulness of highly emotional standardized role-playing sessions with simulators. Psycho-Oncology, 2000. 9(4): p. 293-302.
4. Libert, Y., et al., Predictors of physicians' satisfaction with their management of uncertainty during a decision-making encounter with a simulated advanced stage cancer patient. Patient education and counseling, 2016. 99(7): p. 1121-1129
5. Liénard, A., et al., Is it possible to improve residents breaking bad news skills? A randomised study assessing the efficacy of a communication skills training program. British Journal of Cancer, 2010. 103(2): p. 171-177.
6. Gibon, A.-S., et al., Development of the LaComm 1.0, A French medical communication analysis software: A study assessing its sensitivity to change. Patient Education and Counseling, 2016.
7. Ménard C., et al., Development of the Multi-Dimensional Analysis of Patient Outcome Predictions during Medical Encounters. Patient Education and Counseling, Submitted.
8. Meunier, J., et al., The effect of communication skills training on residents' physiological arousal in a breaking bad news simulated task. Patient Education Counseling, 2013. 93(1): p. 40-7.

ELIGIBILITY:
Inclusion criteria:

* to speak French
* to be willing to participate in the research program
* to be oncologist, other specialist, or resident with at least one year of experience working with cancer patients (part-time or full-time).
* to provide written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Physicians' acquisition of communication skills addressing uncertainty and hope in encounters with a simulated advanced stage cancer patient through validated tools and questionnaires | 4 months

SECONDARY OUTCOMES:
Improvement in physicians satisfaction regarding their communication skills addressing uncertainty and hope in encounters with a simulated advanced stage cancer patient through a questionnaire | 4 months

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Libert Yves, Brussels
  - Libert, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bragard I, Etienne AM, Merckaert I, Libert Y, Razavi D. Efficacy of a communication and stress management training on medical residents' self-efficacy, stress to communicate and burnout: a randomized controlled study. J Health Psychol. 2010 Oct;15(7):1075-81. doi: 10.1177/1359105310361992. Epub 2010 May 7. PMID 20453053
- [Background] Bragard I, Etienne AM, Libert Y, Merckaert I, Lienard A, Meunier J, Delvaux N, Hansez I, Marchal S, Reynaert C, Slachmuylder JL, Razavi D. Predictors and correlates of burnout in residents working with cancer patients. J Cancer Educ. 2010 Mar;25(1):120-6. doi: 10.1007/s13187-010-0050-9. Epub 2010 Feb 26. PMID 20186520
- [Background] Bragard I, Razavi D, Marchal S, Merckaert I, Delvaux N, Libert Y, Reynaert C, Boniver J, Klastersky J, Scalliet P, Etienne AM. Teaching communication and stress management skills to junior physicians dealing with cancer patients: a Belgian Interuniversity Curriculum. Support Care Cancer. 2006 May;14(5):454-61. doi: 10.1007/s00520-005-0008-3. Epub 2006 Jan 18. PMID 16418828
- [Background] Bragard I, Libert Y, Etienne AM, Merckaert I, Delvaux N, Marchal S, Boniver J, Klastersky J, Reynaert C, Scalliet P, Slachmuylder JL, Razavi D. Insight on variables leading to burnout in cancer physicians. J Cancer Educ. 2010 Mar;25(1):109-15. doi: 10.1007/s13187-009-0026-9. PMID 20082173
- [Background] Delvaux N, Merckaert I, Marchal S, Libert Y, Conradt S, Boniver J, Etienne AM, Fontaine O, Janne P, Klastersky J, Melot C, Reynaert C, Scalliet P, Slachmuylder JL, Razavi D. Physicians' communication with a cancer patient and a relative: a randomized study assessing the efficacy of consolidation workshops. Cancer. 2005 Jun 1;103(11):2397-411. doi: 10.1002/cncr.21093. PMID 15858816
- [Background] Gibon AS, Merckaert I, Lienard A, Libert Y, Delvaux N, Marchal S, Etienne AM, Reynaert C, Slachmuylder JL, Scalliet P, Van Houtte P, Coucke P, Salamon E, Razavi D. Is it possible to improve radiotherapy team members' communication skills? A randomized study assessing the efficacy of a 38-h communication skills training program. Radiother Oncol. 2013 Oct;109(1):170-7. doi: 10.1016/j.radonc.2013.08.019. Epub 2013 Sep 7. PMID 24021347
- [Background] Libert Y, Merckaert I, Reynaert C, Delvaux N, Marchal S, Etienne AM, Boniver J, Klastersky J, Scalliet P, Slachmuylder JL, Razavi D. Does psychological characteristic influence physicians' communication styles? Impact of physicians' locus of control on interviews with a cancer patient and a relative. Support Care Cancer. 2006 Mar;14(3):230-42. doi: 10.1007/s00520-005-0871-y. Epub 2005 Jul 29. PMID 16052317
- [Background] Libert Y, Merckaert I, Reynaert C, Delvaux N, Marchal S, Etienne AM, Boniver J, Klastersky J, Scalliet P, Slachmuylder JL, Razavi D. Physicians are different when they learn communication skills: influence of the locus of control. Psychooncology. 2007 Jun;16(6):553-62. doi: 10.1002/pon.1098. PMID 16988932
- [Background] Libert Y, Janne P, Razavi D, Merckaert I, Scalliet P, Delvaux N, Etienne AM, Conradt S, Klastersky J, Boniver J, Reynaert C. Impact of medical specialists' locus of control on communication skills in oncological interviews. Br J Cancer. 2003 Feb 24;88(4):502-9. doi: 10.1038/sj.bjc.6600797. PMID 12592362
- [Background] Lienard A, Merckaert I, Libert Y, Delvaux N, Marchal S, Boniver J, Etienne AM, Klastersky J, Reynaert C, Scalliet P, Slachmuylder JL, Razavi D. Factors that influence cancer patients' anxiety following a medical consultation: impact of a communication skills training programme for physicians. Ann Oncol. 2006 Sep;17(9):1450-8. doi: 10.1093/annonc/mdl142. Epub 2006 Jun 26. PMID 16801333
- [Background] Lienard A, Merckaert I, Libert Y, Delvaux N, Marchal S, Boniver J, Etienne AM, Klastersky J, Reynaert C, Scalliet P, Slachmuylder JL, Razavi D. Factors that influence cancer patients' and relatives' anxiety following a three-person medical consultation: impact of a communication skills training program for physicians. Psychooncology. 2008 May;17(5):488-96. doi: 10.1002/pon.1262. PMID 17879970
- [Background] Lienard A, Merckaert I, Libert Y, Bragard I, Delvaux N, Etienne AM, Marchal S, Meunier J, Reynaert C, Slachmuylder JL, Razavi D. Is it possible to improve residents breaking bad news skills? A randomised study assessing the efficacy of a communication skills training program. Br J Cancer. 2010 Jul 13;103(2):171-7. doi: 10.1038/sj.bjc.6605749. PMID 20628395
- [Background] Lienard A, Merckaert I, Libert Y, Bragard I, Delvaux N, Etienne AM, Marchal S, Meunier J, Reynaert C, Slachmuylder JL, Razavi D. Transfer of communication skills to the workplace during clinical rounds: impact of a program for residents. PLoS One. 2010 Aug 26;5(8):e12426. doi: 10.1371/journal.pone.0012426. PMID 20865055
- [Background] Menard C, Merckaert I, Razavi D, Libert Y. Decision-making in oncology: a selected literature review and some recommendations for the future. Curr Opin Oncol. 2012 Jul;24(4):381-90. doi: 10.1097/CCO.0b013e328354b2f6. PMID 22572724
- [Background] Merckaert I, Lienard A, Libert Y, Bragard I, Delvaux N, Etienne AM, Marchal S, Meunier J, Reynaert C, Slachmuylder JL, Razavi D. Is it possible to improve the breaking bad news skills of residents when a relative is present? A randomised study. Br J Cancer. 2013 Nov 12;109(10):2507-14. doi: 10.1038/bjc.2013.615. Epub 2013 Oct 15. PMID 24129243
- [Background] Merckaert I, Libert Y, Delvaux N, Marchal S, Boniver J, Etienne AM, Klastersky J, Reynaert C, Scalliet P, Slachmuylder JL, Razavi D. Factors influencing physicians' detection of cancer patients' and relatives' distress: can a communication skills training program improve physicians' detection? Psychooncology. 2008 Mar;17(3):260-9. doi: 10.1002/pon.1233. PMID 17575569
- [Background] Merckaert I, Libert Y, Delvaux N, Marchal S, Boniver J, Etienne AM, Klastersky J, Reynaert C, Scalliet P, Slachmuylder JL, Razavi D. Factors that influence physicians' detection of distress in patients with cancer: can a communication skills training program improve physicians' detection? Cancer. 2005 Jul 15;104(2):411-21. doi: 10.1002/cncr.21172. PMID 15952179
- [Background] Meunier J, Merckaert I, Libert Y, Delvaux N, Etienne AM, Lienard A, Bragard I, Marchal S, Reynaert C, Slachmuylder JL, Razavi D. The effect of communication skills training on residents' physiological arousal in a breaking bad news simulated task. Patient Educ Couns. 2013 Oct;93(1):40-7. doi: 10.1016/j.pec.2013.04.020. Epub 2013 May 29. PMID 23726746
- [Background] Meunier J, Libert Y, Merckaert I, Delvaux N, Etienne AM, Lienard A, Marchal S, Reynaert C, Slachmuylder JL, Razavi D. How much is residents' distress detection performance during a clinical round related to their characteristics? Patient Educ Couns. 2011 Nov;85(2):180-7. doi: 10.1016/j.pec.2010.09.022. Epub 2010 Dec 4. PMID 21131159
- [Background] Razavi D, Merckaert I, Marchal S, Libert Y, Conradt S, Boniver J, Etienne AM, Fontaine O, Janne P, Klastersky J, Reynaert C, Scalliet P, Slachmuylder JL, Delvaux N. How to optimize physicians' communication skills in cancer care: results of a randomized study assessing the usefulness of posttraining consolidation workshops. J Clin Oncol. 2003 Aug 15;21(16):3141-9. doi: 10.1200/JCO.2003.08.031. PMID 12915605
- [Background] Razavi D, Delvaux N, Marchal S, De Cock M, Farvacques C, Slachmuylder JL. Testing health care professionals' communication skills: the usefulness of highly emotional standardized role-playing sessions with simulators. Psychooncology. 2000 Jul-Aug;9(4):293-302. doi: 10.1002/1099-1611(200007/08)9:43.0.co;2-j. PMID 10960927
- [Derived] Libert Y, Peternelj L, Bragard I, Lienard A, Merckaert I, Reynaert C, Razavi D. Communication about uncertainty and hope: A randomized controlled trial assessing the efficacy of a communication skills training program for physicians caring for cancer patients. BMC Cancer. 2017 Jul 10;17(1):476. doi: 10.1186/s12885-017-3437-8. PMID 28693515